CLINICAL TRIAL: NCT03339128
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Ranging Study to Evaluate the Safety and Efficacy of Eluxadoline in Pediatric Participants (Age 6 to 17 Years) With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Brief Title: Study to Explore the Therapeutic Effect of Eluxadoline in Treating Irritable Bowel Syndrome With Diarrhea in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3030-202-002; 2017-003770-14 (EudraCT Number)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome with Diarrhea; IBS; IBSD; IBS-D; Irritable Bowel Syndrome; Pediatric
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — eluxadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Eluxadoline 25mg (Experimental): Eluxadoline 25mg, oral administration, twice daily
  Interventions: Drug: Eluxadoline
- Eluxadoline 50mg (Experimental): Eluxadoline 50mg, oral administration, twice daily
  Interventions: Drug: Eluxadoline
- Eluxadoline 100mg (Experimental): Eluxadoline 100mg, oral administration, twice daily
  Interventions: Drug: Eluxadoline
- Placebo (Experimental): Dose-matched placebo, oral administration, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eluxadoline — Oral tablets
  Other Names: Viberzi
  Arms: Eluxadoline 100mg; Eluxadoline 25mg; Eluxadoline 50mg
Drug: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to explore the therapeutic effect of eluxadoline in treating irritable bowel syndrome with diarrhea (IBS-D) in pediatric participants 6-17 years of age, to evaluate the pharmacokinetics of eluxadoline in pediatric participants with IBS-D, and to evaluate the safety and tolerability of eluxadoline in pediatric participants with IBS-D. Enrollment of 12-17 years old age group is closed, enrollment of the 6-11 years old age group will continue.

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide written or verbal informed assent and the parent/guardian/LAR must provide written informed consent before the initiation of any study-specific procedures.
* Participant is a male or female outpatient, 6 to 17 years of age inclusive, at the time the participant provides assent for the study and parent/guardian/LAR has provided signed consent.
* Participant is able to read and understand the assessments in the eDiary. If the participant is 6 to 11 years of age and does not meet this criterion, the interviewer-administered version of the eDiary must be used and the parent/guardian/LAR or caregiver who will be administering the interviewer-administered version of the eDiary must be able to read and understand the assessments in the eDiary and must undergo training.
* Female participants must not be pregnant, breastfeeding, or considering becoming pregnant during the study or for approximately 30 days after the last dose of study drug. Female participants of childbearing potential must have a negative serum pregnancy test at Visit 1 (screening) and a negative urine pregnancy test at Visit 3 (randomization) prior to dosing.
* Female participants of childbearing potential must practice at least 1 protocol-specified method of birth control, that is effective from Study Day 1 through at least 30 days after the last dose of study drug. Local practices may require 2 methods of birth control. Female participants of non-childbearing potential do not need to use birth control.
* Participant has a diagnosis of IBS-D as defined by the modified Rome IV child/adolescent criteria: Must include all of the following:

  -- Abdominal pain at least 4 days per month over at least 2 months associated with one or more of the following:
  * Related to defecation
  * A change in frequency of stool
  * A change in form (appearance) of stool

    * After appropriate evaluation, the symptoms cannot be fully explained by another medical condition.
    * Participant has predominantly diarrheal stool symptoms defined as Bristol stool types 6 or 7 for more than 25% of bowel movements and Bristol stool types 1 or 2 for less than 25% of bowel movements that occur in the absence of laxative.
  * Participant may be newly diagnosed with IBS-D by the investigator at Visit 1. All criteria for diagnosis must be fulfilled for at least 2 months prior to Visit 1 (screening).
* Participant has been compliant with the eDiary by completing both the morning and evening assessments for at least 8 out of the 14 days immediately preceding Visit 3 (randomization).
* Participant has an average daytime abdominal pain score greater than or equal to 1.0 over the 2 weeks prior to randomization.
* Participant has at least 1 daytime bowel movement with a consistency of Type 6 or Type 7 on the pediatric Bristol Stool Form Scale (p-BSFS) on at least 2 days per week during the 2 weeks immediately prior to randomization and that occurs in the absence of laxatives.

Exclusion Criteria:

* Participant has no gallbladder, (ie, agenesis of the gallbladder or cholecystectomy).
* Participant has had any of the following surgeries:

  * Any abdominal surgery within the 3 months prior to Screening; or
  * A history of major gastric, hepatic, pancreatic, or intestinal surgery. (Note: appendectomy, hemorrhoidectomy, or polypectomy greater than 3 months post-surgery are allowed. For the purposes of this study, laparoscopic surgeries without complication are considered minor and non-exclusionary, provided the condition for which the surgery was performed was not exclusionary.)
* Participant has a history of chronic or severe constipation or sequelae from constipation, or known or suspected mechanical GI obstruction or pseudo obstruction.
* Participant has a history or current diagnosis of constipation with encopresis.
* Participant meets the child/adolescent Rome IV criteria of IBS with constipation, IBS with constipation and diarrhea (mixed), unspecified IBS, or functional constipation.
* Participant has a history of intestinal obstruction, stricture, toxic megacolon, GI perforation, fecal impaction, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation.
* Participant has a documented history of hepatic impairment as defined by Child-Pugh Classification Grade A, B or C.
* Participant has a history or current diagnosis of inflammatory or immune-mediated lower GI disorders including inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, microscopic colitis). Crohn's disease affecting the upper GI tract would also be exclusionary.
* Participant has celiac disease, or a positive serological test for celiac disease and the condition has not been ruled out by endoscopic biopsy.
* Participant has any congenital and/or acquired malabsorption syndrome (eg, Shwachman-Diamond syndrome).
* Participant has a history of a microbiologically documented (ie, stool culture or medical history) GI infection within 3 months prior to Screening.
* Participant has a known lactose or fructose intolerance that is associated with diarrhea, abdominal pain or discomfort, and that could confound assessments in the study.
* Participant has a history of diverticulitis within 3 months prior to Screening.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in stool consistency averaged over the 4-week Treatment Period | Baseline (2 Weeks prior to randomization) to Week 4
  Stool consistency will be assessed using the Pediatric Bristol Stool Form Scale (p-BSFS) on a range from 1 (Hard Lumps) to 7 (Watery).

SECONDARY OUTCOMES:
Change from baseline in stool consistency for daily daytime and nighttime stool consistency scores | Baseline (2 Weeks prior to randomization) to Week 4
  Stool consistency will be assessed using the Pediatric Bristol Stool Form Scale (p-BSFS) on a range from 1 (Hard Lumps) to 7 (Watery).
Change from baseline for daytime, nighttime, and 24-hour abdominal pain scores | Baseline (2 Weeks prior to randomization) to Week 4
  Abdominal Pain is scored on a five-point ordinal scale, with 0 meaning no pain, and 4 meaning a lot of pain.
Change from baseline for daytime, nighttime, and 24-hour bowel movement frequency | Baseline (2 Weeks prior to randomization) to Week 4
  Change from baseline in the number of bowel movements.
Change from baseline for daytime, nighttime, and 24 hour urgency-free days | Baseline (2 Weeks prior to randomization) to Week 4
  Change from baseline in the number of urgency free days in a week.
Change from baseline for daytime, nighttime, and 24 hour number of fecal incontinence-free days | Baseline (2 Weeks prior to randomization) to Week 4
  Change from baseline in the number of fecal incontinence-free days in a week.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (46):
- United States (26):
  - HealthStar Research of Hot Springs PLLC /ID# 234609, Hot Springs, Arkansas
  - Applied Research Center of Arkansas /ID# 238070, Little Rock, Arkansas
  - Kindred Medical Institute, LLC /ID# 237368, Corona, California
  - Duplicate_VVCRD Research /ID# 234606, Garden Grove, California
  - Duplicate_Center for Clinical Trials LLC /ID# 234630, Paramount, California
  - Sunrise Research Institute /ID# 237382, Miami, Florida
  - South Miami Medical & Research Group Inc. /ID# 234655, Miami, Florida
  - Valencia Medical & Research Center /ID# 234672, Miami, Florida
  - Florida Research Center, Inc. /ID# 236514, Miami, Florida
  - Duplicate_Wellness Clinical Research /ID# 237401, Miami Lakes, Florida
  - Global Research Associates /ID# 234646, Atlanta, Georgia
  - Children's Ctr Digestive, US /ID# 237575, Atlanta, Georgia
  - Sleep Care Research Institute d/b/a Clinical Research Institute /ID# 236343, Stockbridge, Georgia
  - Advocate Children's Hospital-Park Ridge /ID# 235388, Park Ridge, Illinois
  - Indiana University Health Riley Hospital for Children /ID# 235400, Indianapolis, Indiana
  - Michael W. Simon, MD, PSC /ID# 236517, Lexington, Kentucky
  - Frederick County Pediatrics /ID# 234519, New Market, Maryland
  - MNGI Digestive Health, P. A. /ID# 238057, Minneapolis, Minnesota
  - Celen Medical Group Corp /ID# 234922, Marlton, New Jersey
  - IPS Research Company /ID# 237672, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia - Main /ID# 234313, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Inc. /ID# 236436, Pittsburgh, Pennsylvania
  - Cook Children's Med. Center /ID# 237537, Fort Worth, Texas
  - Texas Children's Hospital /ID# 238304, Houston, Texas
  - Sun Research Institute /ID# 236933, San Antonio, Texas
  - West Virginia University Hospitals /ID# 256841, Morgantown, West Virginia
- Bulgaria (3):
  - Medical center 1 Sevlievo /ID# 237473, Sevlievo, Gabrovo
  - MHATSv.Ivan Rilski /ID# 235399, Kozloduy
  - University Hospital Plovdiv /ID# 235450, Plovdiv
- Canada (2):
  - Duplicate_Edmonton Clinic Health Academy (ECHA) /ID# 234917, Edmonton
  - Manitoba Institute of Child Health /ID# 235448, Winnepeg
- HELIOS Klinikum Wuppertal /ID# 237322, Wuppertal, Germany
- Hungary (3):
  - Eszak-Kozep-budai Centrum, Uj Szent Janos Korhaz /ID# 236993, Budapest
  - Soproni Erzsebet Oktato Korhaz es Rehabilitacios Intezet /ID# 237341, Sopron
  - Vita Verum Medical Bt. /ID# 234321, Székesfehérvár
- Duplicate_Academisch Medisch Centrum /ID# 237117, Amsterdam, North Holland, Netherlands
- Poland (6):
  - Specjalistyczne Gabinety Sp. z o.o. /ID# 236347, Krakow, Lesser Poland Voivodeship
  - Centrum Zdrowia MDM /ID# 237269, Warsaw, Masovian Voivodeship
  - Duplicate_Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 234311, Warsaw, Masovian Voivodeship
  - Korczowski Bartosz Gabinet Lekarski /ID# 234683, Rzeszów, Podkarpackie Voivodeship
  - Copertnicus Podmiot Leczniczy Sp. z o.o. /ID# 235656, Gdansk, Pomeranian Voivodeship
  - Instytut Centrum Zdrowia Matki Polki /ID# 237438, Lodz, Łódź Voivodeship
- Hospital Universitario Dr. Peset /ID# 236755, Valencia, Spain
- United Kingdom (3):
  - Kings College Hospital NHS Foundation Trust /ID# 236305, London, Greater London
  - Duplicate_Manchester University NHS Foundation Trust /ID# 234663, Manchester, Lancashire
  - Blackpool Teaching Hospitals NHS Foundation Trust /ID# 237273, Blackpool

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=3030-202-002